CLINICAL TRIAL: NCT00005958
Title: Treatment of Patients With Transitional-Cell Carcinoma of the Urothelial Tract With Gemcitabine, Docetaxel and Filgrastim
Brief Title: Combination Chemotherapy Plus Filgrastim in Treating Patients With Locally Recurrent or Advanced Urothelium Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amgen (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067939; AMGEN-GCSF-990125; NCI-V00-1594
Record Dates: First submitted 2000-07-05; First posted 2004-04-20 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-10

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter
Keywords: stage III bladder cancer; recurrent bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Filgrastim; Docetaxel; Gemcitabine

INTERVENTIONS:
Biological: filgrastim
Drug: docetaxel
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy with gemcitabine and docetaxel plus filgrastim in treating patients who have locally recurrent or advanced urothelium cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of gemcitabine, docetaxel, and filgrastim (G-CSF) in patients with locally recurrent or advanced transitional cell carcinoma of the urothelial tract. II. Determine the toxicity of this regimen in these patients. III. Determine the disease-free and overall survival of this patient population treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to prior chemotherapy (yes vs no). Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and docetaxel IV over 1 hour on day 8. Patients also receive filgrastim (G-CSF) subcutaneously daily beginning on day 9 and continuing until blood counts recover. Treatment continues every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients who respond to treatment may undergo surgery and 6-8 weeks later receive 2 more courses of chemotherapy. Patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 23-40 patients who have not received prior chemotherapy and 23 patients who have received prior chemotherapy will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven locally recurrent or advanced transitional cell carcinoma (TCC) of the urothelial tract (bladder, renal pelvis, or ureter) or TCC with squamous cell or glandular elements not amenable to curative treatment No pure squamous cell carcinoma or adenocarcinoma Regional or distant metastases after cystoprostatectomy No brain metastases

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: Karnofsky 80-100% Life expectancy: At least 3 months Hematopoietic: No hemorrhagic disorder Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10.0 g/dL Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 3 times ULN Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No known sensitivity to any products to be administered or E. coli derived products No prior other malignancy except inactive nonmelanoma skin cancer, adequately treated stage I or II cancer in complete remission, or early stage prostate cancer (not currently being treated) No illness or psychiatric condition that would preclude study or follow up Not previously entered in this study No active uncontrolled infection

PRIOR CONCURRENT THERAPY: Biologic therapy: No other concurrent biologic therapy No concurrent WBC transfusions Chemotherapy: No prior gemcitabine or docetaxel Other prior chemotherapy allowed Prior intravesical therapy allowed No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy to renal pelvis or ureter allowed Surgery: See Disease Characteristics Cystoprostatectomy or nephroureterectomy for localized TCC allowed Other: No prior investigational drugs No other concurrent investigational therapy No concurrent acetaminophen for fever prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tam, Study Chair — Amgen
Locations (12):
- United States (12):
  - University of California San Diego, La Jolla, California
  - Sacramento Center for Hematology and Medical Oncology, Sacramento, California
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Center for Hematology-Oncology, Boca Raton, Florida
  - Oncology-Hematology Associates of North Illinois, Ltd., Gurnee, Illinois
  - Maine Center for Cancer Medicine and Blood Disorders, Scarborough, Maine
  - St. Joseph Medical Center, Towson, Maryland
  - Hematology & Oncology Associates of Southern Michigan, Jackson, Michigan
  - Hematology Oncology Associates of Central New York, Syracuse, New York
  - Memphis Cancer Center, Inc., Memphis, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - Northern Virginia Oncology Group, Fairfax, Virginia